CLINICAL TRIAL: NCT02595970
Title: A 52-week (Plus Extension Until Commercialization), Single-arm Study to Evaluate Psoriasis Severity and Its Psychosocial Impact Using the Simplified Psoriasis Index (SPI) at 16 Weeks, as Well as Long-term Safety, Tolerability and Efficacy of Secukinumab Administered Subcutaneously in Participants Suffering From Moderate to Severe Psoriasis
Brief Title: Study to Evaluate Psoriasis Severity and Its Psychosocial Impact Using the Simplified Psoriasis Index (SPI), as Well as Long-term Safety, Tolerability and Efficacy of Secukinumab Administered Subcutaneously in Patients With Moderate to Severe Psoriasis
Acronym: IPSI-PSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457AFR01
Record Dates: First submitted 2015-02-25; First posted 2015-11-04 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Secukinumab; Simplified Psoriasis Index; CAIN457A; AIN457AFR01; AIN457A; Skin condition; skin disease; itching condition; psoriasis vulgaris; relapsing/remitting psoriasis; immune-mediated systemic disease; skin lesions; red skin lesions; scaly patches; papules; plaques; itching
MeSH Terms: conditions — Psoriasis; Skin Diseases; Recurrence; Plaque, Amyloid; Pruritus | interventions — secukinumab

STUDY DESIGN:
Masking Description: This was an open label single-arm study; therefore treatment blinding was not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secukinumab (Experimental): Weekly sub cutaneous injections of 300 mg during the first month and then Monthly until Week 52 plus extension until 03/11/2016.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — weekly sub cutaneous injections of 300 mg during the first month and then monthly until week 52 plus extension until 03/11/2016.
  Other Names: open label, no other intervention

SUMMARY:
Evaluate psoriasis severity and its psychosocial impact using a novel Patient Reported Outcome (the Simplified Psoriasis Index SPI) at 16 weeks, as well as long-term safety, tolerability and efficacy of secukinumab administered subcutaneously during 52 weeks (plus extension) in patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
Study to Evaluate Psoriasis Severity and Its Psychosocial Impact Using the Simplified Psoriasis Index (SPI), as Well as Long-term Safety, Tolerability and Efficacy of Secukinumab Administered Subcutaneously in Patients With Moderate to Severe Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of chronic, moderate to severe plaque psoriasis (PASI ≥12; BSA (body surface area) ≥10 and IGA mod 2011 (Investigator's Global Assessment) ≥3) for at least 6 months
* patient candidates for systemic therapy.
* informed consent.

Exclusion Criteria:

* previous treatment with agent targeting IL-17 (interleukine-17) or IL-17 receptor.
* recent treatment with topical treatment (2 weeks), systemic agents (4 weeks for methotrexate, Ciclosporine A; systemic retinoids and other systemic treatment), TNF (tumor necrosis factor) inhibitors (3 months) or IL-12/23 inhibitors (6 months).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PHILIPPE CELERIER, Principal Investigator — HOPITAL SAINT LOUIS - LA ROCHELLE; MARIE-ALETH RICHARD, Principal Investigator — HOPITAL TIMONES - MARSEILLE; SELIM ARACTINGI, Principal Investigator — HOPITAL COCHIN - PARIS; PIERRE ANDRE BECHEREL, Principal Investigator — HOPITAL PRIVE D'ANTONY - ANTONY; EMMANUEL MAHE, Principal Investigator — CH VICTOR DUPOUY - ARGENTEUIL; PHILIPPE LACOUR, Principal Investigator — HOPITAL L'ARCHET - NICE; MIREILLE RUER MULARD, Principal Investigator — CABINET BATEAU BLANC - MARTIGUES; THIERRY BOYE, Principal Investigator — HIA SAINTE ANNE - TOULON; ANNE DUVAL-MODESTE, Principal Investigator — HOPITAL CHARLES NICOLLE - ROUEN; MARIE BEYLOT-BARRY, Principal Investigator — HOPITAL SAINT ANDRE - BORDEAUX; LAURENT MISERY, Principal Investigator — HOPITAL MORVAN - BREST; VINCENT DESCAMPS, Principal Investigator — HOPITAL BICHAT CLAUDE BERNARD - PARIS; GUILLAUME CHABY, Principal Investigator — CHU AMIENS NORD - AMIENS; CARLE PAUL, Principal Investigator — HOPITAL LARREY - TOULOUSE; CHRISTOPHE BEDANE, Principal Investigator — HOPITAL DUPUYTREN - LIMOGES; HERVÉ MAILLARD, Principal Investigator — CENTRE HOSPITALIER LE MANS - LE MANS; JEAN-FRANCOIS CUNY, Principal Investigator — HIA LEGOUEST - METZ
Locations (16):
- France (16):
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study centers: This study involved 17 active centers who enrolled (or recruited) patients in France
  First patient enrolled: 20-May-2015
  Last patient completed: 09-Feb-2017
Pre-assignment Details: No significant events in the study (for example, wash out, run-in) that occur after participant enrollment, but prior to assignment of participants to the treatment arm
Groups:
- Single Arm Secukinumab: Weekly injections of 300mg of secukinumab during the first month (induction period), followed by monthly injections thereafter to week 48. During this extension period, patients continued to receive monthly injections until End of Extension visit.
Period: Overall Study
Arm/Group | Single Arm Secukinumab
Started | 120
Completed | 100 (Out of 100 patients who completed treatment period 2, 20 patients completed the extension period.)
Not Completed | 20
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Not completed — Protocol Violation | 4
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 7

BASELINE CHARACTERISTICS:
Population: FAS
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 116
  More than one race | 0
  Unknown or Not Reported | 0
proSPI (s) [Mean (Standard Deviation); unit: scores on a scale] — proSPI (s) score range is 0 to 50. Higher score means worse condition
  scores on a scale | 24.9 (10.71)
saSPI (s) [Mean (Standard Deviation); unit: score on a scale for each domain of SPI] | 23.5 (10.37)

OUTCOME MEASURES:

1. Primary Outcome: proSPI (s) at Week 16 Compared to Baseline
Description: The primary efficacy outcome of this study evaluates the benefit of secukinumab on the severity of psoriasis based on the SPI. This index comprises 3 components: severity (SPIs), psychosocial (SPIp) and intervention (SPIi) and were evaluated by both health care professional (professional, proSPI) and the patient (self-administered: saSPI). Only the severity components were evaluated for the primary objective: proSPI (s) and saSPI (s). Changes at Week 16 compared to Baseline in patients suffering from moderate to severe plaque psoriasis were analyzed for the purpose of this study.
Time Frame: Week 0 (baseline) to 16 weeks
Population: The primary analysis was performed on the FAS. To assess for robustness of the results, the primary analysis was repeated for the FAS (on observed data).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 119
scores on a scale
  W0 | 24.89 (10.747)
  W16 | 2.34 (6.144)
Statistical Analysis 1: Comparison: Single Arm Secukinumab; Test type: Superiority — adjusted for multiplicity using the Hochberg procedure; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -22.6, 95% CI 2-sided [-24.52 to 20.59], Standard Error of Mean 0.99

2. Secondary Outcome: PASI (Psoriasis Area Severity Index) Score
Description: PASI administered by a professional score range: 0 (no disease) to 72 (maximal disease)
Time Frame: week 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 118
scores on a scale
  W0 | 23.09 (10.541)
  W16 | 2.23 (3.927)
  W52: number analyzed (Participants) | 92
  W52 | 3.16 (5.427)

3. Secondary Outcome: Correlation Between PASI and proSPI (s)
Description: Psoriasis Area Severity Index vs Professional Version of Simplified Psoraisis Index (proSPI) score
Time Frame: week 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Number (95% Confidence Interval); unit: Spearman Correlation coefficient
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 118
Spearman Correlation coefficient
  W0 | 0.691 [0.58 to 0.78]
  W16: number analyzed (Participants) | 109
  W16 | 0.814 [0.74 to 0.87]
  W52: number analyzed (Participants) | 91
  W52 | 0.927 [0.89 to 0.95]

4. Secondary Outcome: proSPI (s, p and i) Over Time
Description: Professional Version of Simplified Psoriasis Index (proSPI)
  SPI for Simplified Psoriasis Index. SPI is composed of 3 domains :
  * s for the severity, min =0 and max=50
  * p for the psychosocial, min=0 and max=10
  * i for the intervention, min = 0 and max = 10 For each domain, high values represented a worse outcome The 3 subscales cannot be combined Please use sore on a scale for the unit of measure
Time Frame: weeks 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 119
scores on a scale
  proSPI (s) - W0 | 24.89 (10.747)
  proSPI (s) - W16: number analyzed (Participants) | 109
  proSPI (s) - W16 | 1.83 (4.427)
  proSPI (s) - W52: number analyzed (Participants) | 91
  proSPI (s) - W52 | 2.93 (6.557)
  proSPI (p) - W0 | 7.80 (1.885)
  proSPI (p) - W16: number analyzed (Participants) | 108
  proSPI (p) - W16 | 1.34 (2.201)
  proSPI (p) - W52: number analyzed (Participants) | 90
  proSPI (p) - W52 | 1.59 (2.341)
  proSPI (i) - W0 | 4.26 (1.924)
  proSPI (i) - W16: number analyzed (Participants) | 110
  proSPI (i) - W16 | 4.78 (1.633)
  proSPI (i) - W52: number analyzed (Participants) | 91
  proSPI (i) - W52 | 4.67 (1.613)

5. Secondary Outcome: saSPI (s, p and i) Over Time
Description: Self-administered Simplified Psoriasis Index (saSPI)
  SPI for Simplified Psoriasis Index. SPI is composed of 3 domains :
  * s for the severity, min =0 and max=50
  * p for the psychosocial, min=0 and max=10
  * i for the intervention, min = 0 and max = 10 For each domain, high values represented a worse outcome The 3 subscales cannot be combined Please use sore on a scale for the unit of measure
Time Frame: weeks 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Mean (Standard Deviation); unit: saSPI score
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 119
saSPI score
  saSPI(s) - W0 | 23.54 (10.412)
  saSPI(s) - W16: number analyzed (Participants) | 108
  saSPI(s) - W16 | 1.80 (4.319)
  saSPI(s) - W52: number analyzed (Participants) | 89
  saSPI(s) - W52 | 2.15 (4.229)
  saSPI(p) - W0 | 8.18 (1.855)
  saSPI(p) - W16: number analyzed (Participants) | 109
  saSPI(p) - W16 | 1.54 (2.299)
  saSPI(p) - W52: number analyzed (Participants) | 90
  saSPI(p) - W52 | 1.47 (2.126)
  saSPI(i) - W0 | 4.34 (1.940)
  saSPI(i) - W16: number analyzed (Participants) | 108
  saSPI(i) - W16 | 4.39 (2.221)
  saSPI(i) - W52: number analyzed (Participants) | 87
  saSPI(i) - W52 | 4.33 (2.276)

6. Secondary Outcome: DLQI (Dermatology Life Quality Index) Over Time
Description: DLQI score has a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired
  MEANING OF DLQI SCORES 0 - 1 no effect on patient's life 2 - 5 small effect on patient's life 6 - 10 moderate effect on patient's life 11 - 20 very large effect on patient's life 21 - 30 extremely large effect on patient's life
Time Frame: weeks 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Mean (Standard Deviation); unit: DLQI score (range : 0 - 30)
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 119
DLQI score (range : 0 - 30)
  WO: number analyzed (Participants) | 118
  WO | 13.6 (7.44)
  W16: number analyzed (Participants) | 109
  W16 | 2.1 (3.67)
  W52: number analyzed (Participants) | 90
  W52 | 1.9 (3.37)

7. Secondary Outcome: Self-administered PASI (SA-PASI)
Description: self-administered PASI (SA-PASI) score
Time Frame: weeks 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Mean (Standard Deviation); unit: saPASI score (range: 0 to 72)
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 118
saPASI score (range: 0 to 72)
  WO | 25.8 (13.55)
  W16: number analyzed (Participants) | 109
  W16 | 2.6 (6.66)
  W52: number analyzed (Participants) | 92
  W52 | 3.3 (7.10)

8. Secondary Outcome: Psoriasis Symptom Diary (PSD) Score
Description: assessment of pain, itching and scaling using the Psoriasis Symptom Diary questionnaire over time
  PSD scores range from 0 to 10, with higher scores indicating a worse condition for each assessment: pain, itching and scaling
Time Frame: weeks 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 119
scores on a scale
  Intensity of pain recorded in PSD- W0 | 5.2 (3.18)
  Intensity of pain recorded in PSD - W16: number analyzed (Participants) | 109
  Intensity of pain recorded in PSD - W16 | 0.9 (2.00)
  Intensity of pain recorded in PSD - W52: number analyzed (Participants) | 91
  Intensity of pain recorded in PSD - W52 | 0.9 (1.78)
  Intensity of itching recorded in PSD - W0 | 6.7 (2.85)
  Intensity of itching recorded in PSD - W16: number analyzed (Participants) | 109
  Intensity of itching recorded in PSD - W16 | 1.3 (2.21)
  Intensity of itching recorded in PSD - W52: number analyzed (Participants) | 91
  Intensity of itching recorded in PSD - W52 | 1.4 (2.11)
  Intensity of scaling recorded in PSD - W0 | 6.5 (2.70)
  Intensity of scaling recorded in PSD - W16: number analyzed (Participants) | 109
  Intensity of scaling recorded in PSD - W16 | 1.0 (1.96)
  Intensity of scaling recorded in PSD - W52: number analyzed (Participants) | 91
  Intensity of scaling recorded in PSD - W52 | 1.3 (2.00)

9. Secondary Outcome: Correlation Between proSPI (for Each Component: s, p and i) and DLQI
Description: Correlation between proSPI (for each component: s, p and i) and DLQI is summarized in table below
Time Frame: weeks 0, 16, 52
Population: Full Analysis Set (observed)
Measure: Number (95% Confidence Interval); unit: Spearman correlation coefficient
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 118
Spearman correlation coefficient
  proSPI (s) and DLQI - W0 | 0.224 [0.04 to 0.39]
  proSPI (s) and DLQI - W16: number analyzed (Participants) | 109
  proSPI (s) and DLQI - W16 | 0.418 [0.25 to 0.56]
  proSPI (s) and DLQI - W52: number analyzed (Participants) | 91
  proSPI (s) and DLQI - W52 | 0.514 [0.34 to 0.65]
  proSPI (p) and DLQI - W0 | 0.494 [0.34 to 0.62]
  proSPI (p) and DLQI - W16: number analyzed (Participants) | 108
  proSPI (p) and DLQI - W16 | 0.671 [0.55 to 0.76]
  proSPI (p) and DLQI - W52: number analyzed (Participants) | 90
  proSPI (p) and DLQI - W52 | 0.757 [0.65 to 0.83]
  proSPI (i) and DLQI - W0 | 0.102 [-0.08 to 0.28]
  proSPI (i) and DLQI - W16: number analyzed (Participants) | 110
  proSPI (i) and DLQI - W16 | 0.016 [-0.17 to 0.20]
  proSPI (i) and DLQI - W52: number analyzed (Participants) | 91
  proSPI (i) and DLQI - W52 | 0.131 [-0.08 to 0.33]

10. Secondary Outcome: Correlation Between proSPI (for Components p and i) and PASI
Description: Correlation between proSPI (p, i) and PASI score by visit (Full Analysis Set (observed)) is summarized in table below
Time Frame: Over time (from Week 0 to Week 52)
Population: Full Analysis Set (observed)
Measure: Number (95% Confidence Interval); unit: Spearman correlation coefficient
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 118
Spearman correlation coefficient
  proSPI (p) and PASI - W0 | 0.173 [-0.01 to 0.34]
  proSPI (p) and PASI - W16: number analyzed (Participants) | 108
  proSPI (p) and PASI - W16 | 0.678 [0.56 to 0.77]
  proSPI (p) and PASI - W52: number analyzed (Participants) | 90
  proSPI (p) and PASI - W52 | 0.749 [0.64 to 0.83]
  proSPI (i) and PASI - W0 | 0.014 [-0.17 to 0.19]
  proSPI (i) and PASI - W16: number analyzed (Participants) | 108
  proSPI (i) and PASI - W16 | 0.105 [-0.08 to 0.29]
  proSPI (i) and PASI - W52: number analyzed (Participants) | 90
  proSPI (i) and PASI - W52 | 0.172 [-0.04 to 0.36]

11. Primary Outcome: Changes of saSPI (s) at Week 16 Compared to Baseline
Description: The primary efficacy objective of the study was to evaluate the benefit of secukinumab on the severity of psoriasis based on the SPI. This index comprises 3 components: severity (SPIs), psychosocial (SPIp) and intervention (SPIi) and were evaluated by both health care professional (professional, proSPI) and the patient (self-administered: saSPI). Only the severity components were evaluated for the primary objective: proSPI (s) and saSPI (s). Changes at Week 16 compared to Baseline in patients suffering from moderate to severe plaque psoriasis were analyzed. proSPI (s) score range is 0 to 50. Higher score means worse condition
Time Frame: Week 0 (baseline) to 16 weeks
Population: Full Analysis Set (FAS): The FAS comprised all patients from the IS who were administered at least one dose of investigational drug with at least one Baseline and one post-baseline SPI evaluation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Single Arm Secukinumab
Number analyzed (Participants) | 118
scores on a scale
  W0 | 23.54 (10.412)
  W16 | 1.99 (4.508)
Statistical Analysis 1: Comparison: Single Arm Secukinumab; Test type: Superiority — adjusted; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -21.6, 95% CI 2-sided [-23.52 to 19.58], Standard Error of Mean 0.99

ADVERSE EVENTS:
Time Frame: baseline to 16 weeks
Groups:
- AIN457 300mg: Listed below are the most frequent treatment emergent adverse events irrespective of causality
Arm/Group | AIN457 300mg
All-Cause Mortality (participants affected / at risk) | 2/120
Serious Adverse Events (participants affected / at risk) | 13/120
Other Adverse Events (participants affected / at risk) | 86/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg (N=120)
Coronary artery occlusion (Cardiac disorders) | 1
Punctate keratitis (Eye disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 1
Face oedema (General disorders) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg (N=120)
Diarrhoea (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 10
Bronchitis (Infections and infestations) | 11
Influenza (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 13
Rhinitis (Infections and infestations) | 11
Viral upper respiratory tract infection (Infections and infestations) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13
Headache (Nervous system disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Psoriasis (Skin and subcutaneous tissue disorders) | 11
Hypertension (Vascular disorders) | 9

LIMITATIONS AND CAVEATS:
The two deaths (i.e.; head injury and lymphoma) were not related to the study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT02595970/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT02595970/SAP_001.pdf